CLINICAL TRIAL: NCT02456870
Title: Aging Subcutaneous Adipose Tissue Response to Overfeeding
Brief Title: Expandability of Aging Adipose Tissue
Acronym: EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-2411
Record Dates: First submitted 2015-04-08; First posted 2015-05-29 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Aging; Obesity
Keywords: Adipose tissue; Overfeeding
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MA (Other): Middle-aged overweight and obese men (age 25-40yr)
  Interventions: Other: Overfeeding
- OA (Other): Older overweight and obese men (age 55-75yr)
  Interventions: Other: Overfeeding

INTERVENTIONS:
Other: Overfeeding — Consumption of 40% excess calories for 7 consecutive days

SUMMARY:
The purpose of this pilot study is to determine whether adipose tissue loses some of its ability to expand in response to overfeeding in older compared to younger men. The investigators hypothesize that the adipose tissue response to overfeeding may be weakened in older when compared to younger men, thereby leading to worsened ectopic storage depots for older men.

DETAILED DESCRIPTION:
This pilot study will begin to address whether adipose tissue biology changes with advancing age. Specifically, we will test whether adipose tissue loses some of its ability to expand in response to overfeeding in older compared to younger men. To test this possibility the Investigators will recruit overweight and mildly obese older (age 55-75y) and younger (age 25-40y) men and collect adipose tissue biopsies before and after 7 days of overfeeding. The investigators will test how well the cells in adipose tissue expand in response to overfeeding and whether this differs between younger and older men.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Aged 25-40y OR 55-75y
* BMI 28-35 kg/m2
* Weight stable (±2kg over past 3 mo)
* Sedentary to moderately active (<3 d/wk of exercise lasting >20min)
* Non-smokers (never used or quit >7yrs prior)

Exclusion Criteria:

* Women
* Currently using hormones, glucose or lipid lowering medication
* Engaged in exercise or diet program
* Currently gaining or losing weight or using weight loss drugs
* Diabetes mellitus (diagnosis, treatment, FBG ≥126 mg/dL)
* Uncontrolled metabolic disorders (e.g., thyroid)

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in adipose-derived stem cell (ASC) differentiation (Delta%oil red O+) | 1 wk of overfeeding
  age-related difference in the ASC differentiation response to overfeeding

SECONDARY OUTCOMES:
Change in ASC proliferation (Delta rate of cell growth) | 1 wk of overfeeding
  age-related difference in the ASC proliferative response to overfeeding
Change in expression of C/EBPalpha, C/EBPbeta, PPARgamma2, SREBP1c, SREBf1a, and Wnt10b (fold-changes in mRNA expression) | 1 wk overfeeding
  age-related difference in the pro-adipogenic response to overfeeding
Change in intramyocellular (IMCL) di-saturated diacylglycerol (DAG) localization (Delta %membrane:cytosol) | 1 week overfeeding
  age-related difference in the IMCL DAG response to overfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Rachael E Van Pelt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Univeristy of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Background] Kim JY, van de Wall E, Laplante M, Azzara A, Trujillo ME, Hofmann SM, Schraw T, Durand JL, Li H, Li G, Jelicks LA, Mehler MF, Hui DY, Deshaies Y, Shulman GI, Schwartz GJ, Scherer PE. Obesity-associated improvements in metabolic profile through expansion of adipose tissue. J Clin Invest. 2007 Sep;117(9):2621-37. doi: 10.1172/JCI31021. PMID 17717599
- [Background] Caso G, McNurlan MA, Mileva I, Zemlyak A, Mynarcik DC, Gelato MC. Peripheral fat loss and decline in adipogenesis in older humans. Metabolism. 2013 Mar;62(3):337-40. doi: 10.1016/j.metabol.2012.08.007. Epub 2012 Sep 19. PMID 22999012
- [Background] Tchoukalova YD, Votruba SB, Tchkonia T, Giorgadze N, Kirkland JL, Jensen MD. Regional differences in cellular mechanisms of adipose tissue gain with overfeeding. Proc Natl Acad Sci U S A. 2010 Oct 19;107(42):18226-31. doi: 10.1073/pnas.1005259107. Epub 2010 Oct 4. PMID 20921416